CLINICAL TRIAL: NCT01362569
Title: Endotoxin, Neutrophil Function and Albumin in Renal Insufficiency
Acronym: ENARI
Status: Completed | Type: Observational
Sponsor: Vanessa Stadlbauer-Koellner, MD (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor-Investigator, Vanessa Stadlbauer-Koellner, MD, PD. Dr. med, Medical University of Graz
Organization: Medical University of Graz (Other)
Other Study IDs: P23532
Record Dates: First submitted 2011-05-23; First posted 2011-05-30 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Chronic Renal Insufficiency; Acute Renal Failure
Keywords: endotoxin; neutrophil function; albumin function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- predialytic renal insufficiency: Patents without renal replacement therapy
- hemodialysis/hemofiltration patients: patients undergoing regular hemodialysis/hemofiltration
- peritoneal dialysis patients: patients undergoing peritoneal dialysis
- acute renal failure: patients with acute renal failure
- post renal transplantation: patients after renal transplantation
- healthy controls: control group

SUMMARY:
Chronic kidney disease is widespread in the western world with bacterial infection and sepsis as common complication. It has been shown that innate immune defence, represented by dysfunction of neutrophil granulocytes, is impaired in chronic kidney disease. Another impact of chronic kidney disease on innate immunity is the chronic activation of neutrophils leading to high levels of inflammatory cytokines, thus contributing to protein oxidation. Oxidation of human serum albumin (HSA), the major plasma protein, occurs in chronic kidney disease and leads to further activation of neutrophils. Another important impact of HSA oxidation is the decrease of its binding capacity leading to impaired detoxification ability of albumin. This includes reduced clearance of endotoxin, a major component of the gram negative bacterial cell wall. Circulating endotoxin is recognized by complex formation with lipopolysaccharide binding protein (LBP) followed by binding to CD14 and toll-like receptor (TLR) 4. High systemic endotoxin levels occur in chronic kidney disease and may be the result of decreased clearance ability of HSA and increased gut permeability in combination with intestinal bacterial overgrowth. High systemic endotoxin is associated with worse outcome in several diseases and could be used as predictor for mortality in chronic kidney disease patients.

Endotoxemia in renal insufficiency leads to impaired neutrophil function and to increased albumin oxidation. Oxidized albumin is not able to bind endotoxin adequately any more, which leads to a further increase in oxidative stress and neutrophil dysfunction, resulting in a vicious cycle.

195 patients with renal dysfunction will be enrolled and divided into 5 groups. Additionally, samples of 25 age and sex-matched healthy controls will be collected.

This concept will change the understanding of several aspects of chronic kidney disease and will potentially help to stratify patients into different groups at risk according to their endotoxin status, and their immune and albumin dysfunction. The results of this study will have important implications into the development of novel therapeutic strategies

DETAILED DESCRIPTION:
Laboratory methods Endotoxin will be detected by an adapted limulus amoebocyte lysate assay. LBP and sCD14 will be determined by means of ELISA. HPLC will be used to determine nitrate, nitrite, albumin fractions, albumin binding capacity, iNOS expression and energy status of neutrophils. For investigation of oxidation driven by leukocyte derived myeloperoxidase, mass spectrometry analysis will be used. Carbonyl contents of proteins will be detected by ELISA. Neutrophil function and TLR2, 4 and 9 expression will be studied by flow cytometrical analysis. For cell culture tests, freshly isolated neutrophils or differentiated HL60 cells will be used and incubated with albumin and/or endotoxin. Stool samples will be used for 16srDNA sequencing of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

Age between 18-80 years, informed consent Groups 1a, 1b, 2a, 2b, 3a, 3b Patients with chronic kidney disease as defined previously [65] either

1a) with an eGFR between 30 and 45 (KDIGO 3B)

1. b) with an eGFR between 15 and 30 (KDIGO 4)
2. a) undergoing hemodialysis for ESRD

2b) undergoing hemodiafiltration for ESRD

3a) undergoing peritoneal dialysis for ESRD without signs of infection

3b) undergoing peritoneal dialysis for ESRD with peritonitis ≥2 out of the 4 criteria (>100 leucocytes/50%neutrophils, cloudy peritoneal dialysate, typical clinical presentation with fever and abdominal pain, positive culture from the peritoneal dialysate)

Group 4 Patients with acute kidney injury (AKIN 3 [66] defined as an increase in serum creatinine to 300% (3-fold) from baseline or serum creatinine 4.0 mg/dl with an acute rise of at least 0.5mg/dl or urine output of < 0.3ml/kg/h 24h or anuria 12h) Initiation of acute renal replacement therapy

Group 5 Stable patients after kidney transplantation with either an eGFR > 45, between 30 and 45 or < 30

Group 6: Healthy controls

Exclusion Criteria:

* Malignancy, pregnancy,chronic inflammatory bowel disease, celiac disease, active alcohol abuse, any severe organ dysfunction unrelated to renal dysfunction Groups 1a, 1b, 2a, 2b, 3 Organ transplantation Clinical evidence of active infection (except for group 3b) Treatment with antibiotics within the last 2 weeks (except for group 3b)

Group 4 Preexisting ESRD

Group 5 Clinical evidence of active infection Treatment with antibiotics within the last 2 weeks

Group 6:

Any evidence of acute or chronic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 50 predialytic patients (a) 25 patients with an eGFR between 30 and 45 (KDIGO 3B) and (b) 25 patients with an eGFR between 15 and 30 (KDIGO 4)
  2. 50 patients undergoing hemodialysis or hemodiafiltration for ESRD (a) 25 patients under therapy with sevelamer and (b) 25 patients without sevelamer
  3. (a) 25 patients undergoing peritoneal dialysis for ESRD without signs of infection and (b) 25 patients undergoing peritoneal dialysis for ESRD with peritonitis
  4. 25 patients with acute renal failure
  5. 45 patients after kidney transplantation (a) 15 patients with an eGFR > 45, (b) 15 patients with an eGFR between 30 and 45 and (c) 15 patients with an eGFR < 30
  6. 25 age and sex-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Endotoxin levels (EU/ml and qualitative positive/negative) | Day 0
  Percentage of patients with measurable endotoxin serum levels in each group.

SECONDARY OUTCOMES:
albumin oxidation (%), albumin binding capacity (ratio), neutrophil function (%), | Day 0
  We want to investigate the following in patients with different stages of chronic renal insufficiency.
  Albumin oxidation and function in correlation with the endotoxin status Endotoxin binding to albumin Neutrophil function, energy status and NO metabolism in correlation with the endotoxin status
microbiome composition | Day 0
  In a subgroup of patients undergoing hemodialysis or peritoneal dialysis we will assess the composition of the gut micro biome in stool samples by 16s rDNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Medical Univeristy of Graz
Locations (1):
- Department of Internal Medicine, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided